CLINICAL TRIAL: NCT06413199
Title: Adaptive Response of Brain Towards Resistance Training in Healthy Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Society for Rehabilitation of Differently Abled Hospital (Other)
Collaborators: University of Karachi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSRDHospital
Record Dates: First submitted 2023-10-31; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Resistance Training
Keywords: Resistance Training; Performance; Nervous Response; Muscle growth; Exercise Induced Performance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyper Training Group (Experimental): 2 training session per week for 2 months, 1 set of 10 unloaded repetitions in arms as a warm-up, 4 sets with a goal of 8-12 repetitions with 90 seconds of rest between sets and elbows had to be fully locked out to be counted as a repetition, 1.5 seconds for concentric and 1.5 seconds for eccentric portion.
  Interventions: Other: Hyper Training
- 1 Repetition Maximum Group (Active Comparator): 2 training session per week for 2 months, 1 set of 10 unloaded repetitions in arms as a warm-up, training protocol consisted of 5 attempts to lift as much weight as possible one time for that training visit with 90 seconds of rest between attempts. The load was progressively increased each attempt to try to reach or exceed their previous 1RM.
  Interventions: Other: 1 Repetition maximum training group

INTERVENTIONS:
Other: Hyper Training — Experimental group will perform 2 training session per week for 2 months, 1 set of 10 unloaded repetitions in arms as a warm-up, 4 sets with a goal of 8-12 Reps with 90 seconds rest between sets. 1.5 second concentric and 1.5 second eccentric contraction of bench press, The elbows had to be fully locked out to be counted as a repetition.
  Arms: Hyper Training Group
Other: 1 Repetition maximum training group — 2 training session per week for 8 weeks, 1 set of 10 unloaded repetitions in arms as a warm-up, 1 Repetition maximum training group consisted of 5 attempts to lift as much weight as possible one time for that training visit with 90 seconds of rest between attempts, the load was progressively increased each attempt to try to reach or exceed their previous 1 repetition maximum.
  Arms: 1 Repetition Maximum Group

SUMMARY:
The novelty of this study is to identify the mechanism of nervous system by applying resistance training intervention in healthy individuals.

DETAILED DESCRIPTION:
Resistance training is a form of exercise that is popular particularly for its role in improving athletic performance by increasing muscular strength, power and speed, hypertrophy, local muscular endurance, motor performance, balance and coordination. The objective of the study is to find out the effects of resistance training on Central and Peripheral Nervous System in healthy individuals. A total of 100 participants will be included in the study including both male and female. The study will be divided into two main groups. Experimental group will perform 8-12 Reps with 1.5 sec concentric and 1.5 sec eccentric contraction of bench press with 90 sec of rest between sets with 2 sets per week for 2 months.

1RM of control group will be calculated through the same method and the training protocol for the Control group consisted of 5 attempts to lift as much weight as possible one time for that training visit with 90 seconds of rest between attempts. The load was progressively increased each attempt to try to reach or exceed their previous 1RM.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index should be 18.5-24.9 kg/m2.
* Participants were untrained and had not engaged in resistance exercise within 6 months prior to beginning the study.

Exclusion Criteria:

* Participants with any kind of Gastrointestinal Tract disturbance will be excluded from the study.
* Participants with any kind of Musculoskeletal injury will be excluded from the study.
* Participant with any kind of Neurological disturbance will be excluded from the study.
* Participants who use tobacco products within the previous 6 months.
* Participants who take any type of medication within the previous 6 months.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2024-12-29 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
NCS (Motor Nerve Conduction Study) | • 0 week • 8th week
  To determine how fast or slow the nerves are conducting an electrical current using F wave
EEG (Electroencephalography) | • 0 week • 8th week
  To measure the electrical activity of the brain using alpha and beta waves
Dynamometer | • 0 week • 4th week • 8th week
  To measure the strength after resistance training
Estimation of Albumin & Globulin ratio | • 0 week • 8th week
  To measure the total amount of protein in blood and effects of resistance training

CONTACTS AND LOCATIONS:
Overall Officials: Danish Latif, PhD*, Principal Investigator — PSRD College of Rehabilitation Sciences
Locations (1):
- PSRD Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Comfort P, Haigh A, Matthews MJ. Are changes in maximal squat strength during preseason training reflected in changes in sprint performance in rugby league players? J Strength Cond Res. 2012 Mar;26(3):772-6. doi: 10.1519/JSC.0b013e31822a5cbf. PMID 22310512
- [Background] Brooks JH, Fuller CW, Kemp SP, Reddin DB. Incidence, risk, and prevention of hamstring muscle injuries in professional rugby union. Am J Sports Med. 2006 Aug;34(8):1297-306. doi: 10.1177/0363546505286022. Epub 2006 Feb 21. PMID 16493170
- [Background] Kristensen J, Franklyn-Miller A. Resistance training in musculoskeletal rehabilitation: a systematic review. Br J Sports Med. 2012 Aug;46(10):719-26. doi: 10.1136/bjsm.2010.079376. Epub 2011 Jul 26. PMID 21791457
- [Background] Hakkinen K, Alen M, Komi PV. Changes in isometric force- and relaxation-time, electromyographic and muscle fibre characteristics of human skeletal muscle during strength training and detraining. Acta Physiol Scand. 1985 Dec;125(4):573-85. doi: 10.1111/j.1748-1716.1985.tb07760.x. PMID 4091001
- [Background] Mitchell CJ, Churchward-Venne TA, West DW, Burd NA, Breen L, Baker SK, Phillips SM. Resistance exercise load does not determine training-mediated hypertrophic gains in young men. J Appl Physiol (1985). 2012 Jul;113(1):71-7. doi: 10.1152/japplphysiol.00307.2012. Epub 2012 Apr 19. PMID 22518835
- [Background] Taber CB, Vigotsky A, Nuckols G, Haun CT. Exercise-Induced Myofibrillar Hypertrophy is a Contributory Cause of Gains in Muscle Strength. Sports Med. 2019 Jul;49(7):993-997. doi: 10.1007/s40279-019-01107-8. No abstract available. PMID 31016546
- [Background] Deumens R, Bozkurt A, Meek MF, Marcus MA, Joosten EA, Weis J, Brook GA. Repairing injured peripheral nerves: Bridging the gap. Prog Neurobiol. 2010 Nov;92(3):245-76. doi: 10.1016/j.pneurobio.2010.10.002. Epub 2010 Oct 13. PMID 20950667
- [Background] Dankel SJ, Counts BR, Barnett BE, Buckner SL, Abe T, Loenneke JP. Muscle adaptations following 21 consecutive days of strength test familiarization compared with traditional training. Muscle Nerve. 2017 Aug;56(2):307-314. doi: 10.1002/mus.25488. Epub 2017 Mar 3. PMID 27875635
- [Background] Mattocks KT, Buckner SL, Jessee MB, Dankel SJ, Mouser JG, Loenneke JP. Practicing the Test Produces Strength Equivalent to Higher Volume Training. Med Sci Sports Exerc. 2017 Sep;49(9):1945-1954. doi: 10.1249/MSS.0000000000001300. PMID 28463902
- [Background] Kacin A, Strazar K. Frequent low-load ischemic resistance exercise to failure enhances muscle oxygen delivery and endurance capacity. Scand J Med Sci Sports. 2011 Dec;21(6):e231-41. doi: 10.1111/j.1600-0838.2010.01260.x. Epub 2011 Mar 8. PMID 21385216
- [Background] Jessee MB, Buckner SL, Mouser JG, Mattocks KT, Dankel SJ, Abe T, Bell ZW, Bentley JP, Loenneke JP. Muscle Adaptations to High-Load Training and Very Low-Load Training With and Without Blood Flow Restriction. Front Physiol. 2018 Oct 16;9:1448. doi: 10.3389/fphys.2018.01448. eCollection 2018. PMID 30386254
- [Background] Andersen LL, Andersen JL, Zebis MK, Aagaard P. Early and late rate of force development: differential adaptive responses to resistance training? Scand J Med Sci Sports. 2010 Feb;20(1):e162-9. doi: 10.1111/j.1600-0838.2009.00933.x. Epub 2009 May 26. PMID 19793220
- [Background] Bickel CS, Cross JM, Bamman MM. Exercise dosing to retain resistance training adaptations in young and older adults. Med Sci Sports Exerc. 2011 Jul;43(7):1177-87. doi: 10.1249/MSS.0b013e318207c15d. PMID 21131862
- [Background] Dankel SJ, Kang M, Abe T, Loenneke JP. Resistance training induced changes in strength and specific force at the fiber and whole muscle level: a meta-analysis. Eur J Appl Physiol. 2019 Jan;119(1):265-278. doi: 10.1007/s00421-018-4022-9. Epub 2018 Oct 24. PMID 30357517
- [Background] Griffin L, Cafarelli E. Transcranial magnetic stimulation during resistance training of the tibialis anterior muscle. J Electromyogr Kinesiol. 2007 Aug;17(4):446-52. doi: 10.1016/j.jelekin.2006.05.001. Epub 2006 Aug 7. PMID 16891123
- [Background] Aagaard P, Simonsen EB, Andersen JL, Magnusson P, Dyhre-Poulsen P. Neural adaptation to resistance training: changes in evoked V-wave and H-reflex responses. J Appl Physiol (1985). 2002 Jun;92(6):2309-18. doi: 10.1152/japplphysiol.01185.2001. PMID 12015341
- [Background] Krutki P, Mrowczynski W, Baczyk M, Lochynski D, Celichowski J. Adaptations of motoneuron properties after weight-lifting training in rats. J Appl Physiol (1985). 2017 Sep 1;123(3):664-673. doi: 10.1152/japplphysiol.00121.2017. Epub 2017 Jun 8. PMID 28596267
- [Background] Canepari M, Rossi R, Pellegrino MA, Orrell RW, Cobbold M, Harridge S, Bottinelli R. Effects of resistance training on myosin function studied by the in vitro motility assay in young and older men. J Appl Physiol (1985). 2005 Jun;98(6):2390-5. doi: 10.1152/japplphysiol.01103.2004. Epub 2005 Jan 27. PMID 15677736
- [Background] Chin ER, Olson EN, Richardson JA, Yang Q, Humphries C, Shelton JM, Wu H, Zhu W, Bassel-Duby R, Williams RS. A calcineurin-dependent transcriptional pathway controls skeletal muscle fiber type. Genes Dev. 1998 Aug 15;12(16):2499-509. doi: 10.1101/gad.12.16.2499. PMID 9716403
- [Background] Westerblad H, Allen DG. Changes of myoplasmic calcium concentration during fatigue in single mouse muscle fibers. J Gen Physiol. 1991 Sep;98(3):615-35. doi: 10.1085/jgp.98.3.615. PMID 1761971
- [Background] Coelho HJ Junior, Rodrigues B, de Oliveira Goncalves I, Uchida MC. Effects of a short-term detraining period on muscle functionality and cognition of strength-trained older women: a preliminary report. J Exerc Rehabil. 2017 Oct 30;13(5):559-567. doi: 10.12965/jer.1735010.505. eCollection 2017 Oct. PMID 29114531
- [Background] Ribeiro AS, Tomeleri CM, Souza MF, Pina FL, Schoenfeld BJ, Nascimento MA, Venturini D, Barbosa DS, Cyrino ES. Effect of resistance training on C-reactive protein, blood glucose and lipid profile in older women with differing levels of RT experience. Age (Dordr). 2015 Dec;37(6):109. doi: 10.1007/s11357-015-9849-y. Epub 2015 Oct 26. PMID 26499819